CLINICAL TRIAL: NCT03701035
Title: Does Moderate Intensity Aerobic Training Influence Serum Levels of BDNF in Sub-acute and Chronic Stroke Patients and Consequently Increase the Efficacy of Upper-limb Rehabilitation? A Study Protocol for a Randomized Control Trial With an Embedded Health Economic Evaluation.
Brief Title: Moderate Intensity Aerobic Training in Sub-acute and Chronic Stroke Patients - the Influence on Brain Derived Neurotrophic Factor (BDNF) and Upper-limb Rehabilitation. A Protocol for a Randomized Control Trial and Health Economic Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clare Maguire (Other)
Collaborators: Bildungszetrum Gesundheit Basel-Stadt (Unknown); Rehab Basel (Other)
Responsible Party: Sponsor-Investigator, Clare Maguire, Head of Master Programme Neurorehabilitation, Technical University of Bern
Organization: Technical University of Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-01249
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training & UL Motor Training (Experimental): Aerobic training at 40%-59% Heart Rate Reserve (AT) increasing from personal maximum time (if < 40 mins) to 40 minutes followed by UL motor training with the Armeo®Spring/Senso/Pablo X2® 3 * weekly, 12 weeks
  Interventions: Behavioral: Aerobic Training & UL Motor Training
- Non-aerobic Training & UL Motor Training (Active Comparator): 40 minutes non-aerobic gait & balance circuit training followed by UL motor training with the Armeo®Spring/Senso/Pablo X2® 3 * weekly, 12 weeks
  Interventions: Behavioral: Non-aerobic training & UL Motor Training

INTERVENTIONS:
Behavioral: Aerobic Training & UL Motor Training — Aerobic training at 40%-59% Heart Rate Reserve (AT) increasing from personal maximum time (if < 40 mins) to 40 minutes followed by UL motor training with the Armeo®Spring/Senso/Pablo X2®
  Arms: Aerobic Training & UL Motor Training
Behavioral: Non-aerobic training & UL Motor Training — 40 minutes non-aerobic gait & balance circuit training followed by UL motor training with the Armeo®Spring/Senso/Pablo X2®
  Arms: Non-aerobic Training & UL Motor Training

SUMMARY:
The aim of this study is to evaluate the influence on three different training modalities on the blood concentration levels of a growth factor called Brain Derived Neurotrophic Factor (BDNF) and on the recovery of arm function following in sub-acute and chronic stroke survivors. The training modalities are 1. moderate intensity aerobic training on a bike ergonometer followed by robotic or sensor-based upper-limb training, 2. non-aerobic circuit training followed by robotic or sensor-based upper-limb training 3. circuit training alone.

DETAILED DESCRIPTION:
Background and Rationale:Brain-derived neurotrophic factor (BDNF) belongs to a group of neurotrophins which influence neuroplasticity by increasing long-term potentiation and axonal and dendritic growth. Levels of serum BDNF are increased following moderate intensity aerobic exercise (MAE) in animal and healthy subjects. The influence of MAE on BDNF following stroke and the resultant efficacy of motor training in this environment remains unclear.

Objective(s):To investigate the influence of MAE on acute and chronic levels of serum BDNF in sub-acute and chronic stroke patients, the efficacy of robotic upper limb or sensor based motor task training in this environment and consequent effect on functional arm recovery compared to the same upper limb training following non-aerobic training circuit training, or non-aerobic circuit training alone To evaluate the cost-effectiveness of the interventions. Study Interventions: Group 1: moderate intensity AE 40 minutes, 3 times weekly followed after 20 minutes break by 40 minutes robotic or sensor-based upper-limb Training. Group2: non-aerobic gait and balance circuit training 40 mins 3 times weekly followed after 20 minutes break by 40 minutes robotic or sensor-based upper-limb training, group 3: 40 minutes non-aerobic gait and balance circuit training.In total 45 participants will be enrolled - 15 in each group.Study Duration:3 monthly Intervention period per intervention group, with a 3 month and 6 month follow-up. .

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke ischemic or intracerebral hemorrhagic > 3 months post- stroke
* Active shoulder abduction, wrist and finger extension 10 degrees from a flexed position

Exclusion Criteria:

* Contraindications to maximal exercise testing according to the American College of Sports Medicine guidelines
* Severe perceptual problems
* Concurrent neurological diagnoses e.g. Parkinsons disease
* Comorbidities which may interfere with exercise participation
* Significant cognitive impairment < 24 on the Montreal Cognitive Assessment Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
BDNF | 12 weeks
  Acute (immediate post exercise) and chronic (post-intervention) serum BDNF levels
Action Research Arm Test (ARAT) | 12 weeks
  A 19-Item standardised assessment of UL function measuring ADLs, coordination & dexterity.

SECONDARY OUTCOMES:
The Fugl-Meyer Assessment - Upper Extremity Scale (FMA). | 12 weeks
  Instrument for measuring upper limb impairment after stroke. The Fugl-Meyer Assessment - Upper Extremity Scale (FMA). This is reliable, responsive and valid instrument for measuring upper limb impairment after stroke. Items are scored on a three-point ordinal scale: 0=cannot perform, 1=performs partially, 2=performs fully. Maximal Score 66.
10 meter walking test | 12 weeks
  A measurement of gait speed
Trunk Sway in standing with eyes closed | 12 weeks
  Standing balance
The Montreal Cognitive Assessment (MoCA©). | 12 weeks
  This is a rapid screen of cognitive performance to detect mild cognitive dysfunction. The test consists of 16 items and 11 categories to assess multiple cognitive domains. The maximal score is 30.
Corsi Block Test | 12 weeks
  Evaluates visuospatial short-term working memory
The Fatigue Severity Scale (FSS) | 12 weeks
  Measures post-stroke-fatigue. This is a 9-item, 7 point linkert scale scale which measures the effect of fatigue on activities and lifestyle. The higher the score the worse the fatigue.
Stroke Impact Scale | 12 weeks
  A disease specific Quality of Life measure.This is a 59 item measure in which 8 domains are assessed. Each item is a 5-point Linkert scale related to difficulty completing the scale . Summative scores are generated for each domain. A higher score indicates a better Performance.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Maguire, PhD, Principal Investigator — Bern University of Applied Sciences
Locations (1):
- RehaB clinic for Neurorehabilitation and Paraplegiology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided